CLINICAL TRIAL: NCT05503238
Title: The Effects of Mother-infant Skin-to-skin Contact on Cumulative Stress of Preterm Infants in the Neonatal Intensive Care Unit : A Randomized Controlled Trial
Brief Title: The Effects of Mother-infant Skin-to-skin Contact on Stress Response of Preterm Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The researcher in charge has left the affiliation.
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022 -31
Record Dates: First submitted 2022-07-31; First posted 2022-08-16 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Preterm Infant
Keywords: Stress response; Skin-to-skin contact; Cortisol
MeSH Terms: conditions — Premature Birth; Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin-to-skin contact group (Experimental): Provide maternal-infant skin-to-skin contact for preterm infants in the neonatal intensive care unit.
  Interventions: Behavioral: Skin-to-skin contact; Other: Routine care
- Routine care group (Other): Perform routine nursing care for preterm infants in the neonatal intensive care unit.
  Interventions: Other: Routine care

INTERVENTIONS:
Behavioral: Skin-to-skin contact — Preterm infants will receive maternal-infant skin-to-skin contact at least 1 continuous hour everyday from infant 3 days of life until discharge, and other nursing care will be same as the routine group. During skin-to-skin contact, place naked baby only with diaper on the mother's bare chest in an upright position and tilt the baby's head to one side in a slightly extended position to keeps the airway open, cover the infant with a blanket to keep them warm. A neonatal nurse will be stay with mother and infant to observe and support.
  Arms: Skin-to-skin contact group
Other: Routine care — Preterm infants will receive standard nursing care provided by neonatal nurses in accordance with hospital principles during hospitalization.

SUMMARY:
This study will evaluate the effect of maternal-infant skin-to-skin contact (SSC) versus routine care on general stress in preterm infants in the neonatal intensive care unit (NICU).

DETAILED DESCRIPTION:
Primary outcome of this trial to investigate the effects daily skin-to-skin contact on cumulative stress through measures salivary cortisol. The intervention group will receive mother-infant skin-to-skin contact at least 1 continuous hour everyday from infant 3 days of life until discharge. The control group will receive routine neonatal care during hospitalization except skin-to-skin contact. The concentration of salivary cortisol and other infant and parental outcomes will be measured in both groups.

ELIGIBILITY:
Inclusion Criteria:

* 31 weeks≤gestational age<37 weeks;
* Birth weight ≥ 1500g;
* Admission age < 24h;
* No congenital malformations;
* Vital signs are stable and does not use ventilator and other auxiliary life support systems.

Exclusion Criteria:

* Severe periventricular / intraventricular hemorrhage (grade III);
* Receiving sedation or vasopressor or analgesics opiodis and corticosteroids;
* Mother unable to communicate and communicate normally; Mother has a history of depression.

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes on the concentration of cortisol of preterm infants | From 3 days of life (baseline) to 7 days of life
  At 3 days of life (baseline) and 7 days of life, the saliva sample will collected from preterm infants by a neonatal nurse. The concentration of salivary cortisol will be measured using by radioimmunoassay.

SECONDARY OUTCOMES:
Changes on the level of cortisol during heel lancet | At the preterm infants 7 days of life
  At 7 days of life, saliva sample will collected from preterm infants by a neonatal nurse before and 30 mins after heel lancet.
Score of Edinburgh Postnatal Depression Scale | Through study completion, an average of 40 days
  Mothers' depression status will be measure by Edinburgh Postnatal Depression Scale through WeChat at discharge day. The questionnaire is a self screening tool, contains 10 items, each item is scored from 0-3 according to a 4-point Likert scale , and the total score is 0-30 points. The higher the score, the more severe the depression. All the questionnaires will collect and calculate by a neonatal nurse.
Length of hospital stays | Through study completion, an average of 40 days
  Duration of hospitalization will calculate from the date of admission to the date of discharge, which obtained from clinical records files.
Crying time | At the preterm infants 7 days of life
  At 7 days of life, crying time will be recorded and calculated by a neonatal nurse during heel lancet.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Hu, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No